CLINICAL TRIAL: NCT00345527
Title: A Randomized Control Trial Examining Two Treatments for Problem Gambling
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study moved to British Columbia
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Lorne Korman, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 004/2006
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Gambling, Pathological; Anger
Keywords: Problem gambling; Clinically significant anger
MeSH Terms: conditions — Gambling | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Emotion and Behaviour Regulation Treatment (EBRT)
Behavioral: Cognitive Behavioural Therapy

SUMMARY:
Despite evidence of high rates of concurrent substance use and anger problems among problem gamblers, until recently there have been no empirically evaluated treatments for these co-morbid problems. A recent study (Korman, Collins, McMain, & Skinner, 2005) found that an emotion and behaviour regulation treatment (EBRT) was more effective than a gambling-only treatment-as-usual in engaging clients in treatment and in reducing gambling, anger, and substance use. This study is a replication of Korman et al's study and will compare an emotion and behaviour regulation treatment (EBRT) for problem gambling, anger and substance use to a manualized cognitive behavioural treatment (CBT) for problem gambling.

DETAILED DESCRIPTION:
80 participants will be randomly assigned to either an emotion and behaviour regulation treatment (EBRT) or to a cognitive behavioural treatment (CBT). Randomization will be stratified by the presence of substance dependence disorder. Both treatment conditions will consist of 12 one-hour weekly outpatient individual sessions. Participants will be assessed at baseline, end of treatment, and 3-months, 6-months and 12-months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Problem gambling (PGSI > 7; c.f., Ferris & Wynne, 2001)
* Clinically significant anger (STAXI-II anger expression/trait subscale score >75th percentile and/or Anger Control subscale score < 25th percentile; c.f., Spielberger, 1999)

Exclusion Criteria:

* Major thought disorders
* Acute manic episode
* High psychopathy
* Severe developmental/cognitive disability
* Outstanding legal charges/sentencing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Treatment Retention
The Working Alliance Inventory - Client version (WAI-C)
Canadian Problem Gambling Inventory(CPGI)
State-Trait Anger Expression Inventory-II(STAXI-II)
Addiction Severity Index: Drug and Alcohol Use section
Structured Clinical Interview for the DSM-IV (SCID; APA, 1994), substance use section

CONTACTS AND LOCATIONS:
Overall Officials: Lorne Korman, PhD, Principal Investigator — BC Mental Health and Addiction Services